CLINICAL TRIAL: NCT02170779
Title: Developing and Testing a Comprehensive MS Spasticity Management Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N1401-P
Record Dates: First submitted 2014-06-09; First posted 2014-06-23 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Multiple Sclerosis; Spasticity
Keywords: multiple sclerosis; spasticity; stretching; exercise; rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Spasticity: Take Control (Experimental): 4 visits: baseline, view and discuss DVDs, practice stretching, outcome measures
  Interventions: Behavioral: Spasticity: Take Control
- B Usual care (Other): 2 visits: baseline and given usual treatment of brochure for stretching, outcome measures
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Spasticity: Take Control — 4 visits: baseline, view and discuss DVDs, practice stretching, outcome measures
  Arms: A Spasticity: Take Control
Other: Usual care — 2 visits: baseline followed by usual care of brochure for stretching then outcome measures
  Arms: B Usual care

SUMMARY:
This is a study to determine the impact of education and specific lower extremity stretches for MS-related spasticity. The study will evaluate the acceptance and efficacy of education and stretching using a randomized controlled pilot trial.

DETAILED DESCRIPTION:
Participants have 2-4 visits depending on program assignment. All participants will have screening/baseline and follow-up visits. Participants in the intervention program will have 2 additional visits with a group of other people with MS to view and discuss the DVDs on spasticity education and stretching for lower extremity MS spasticity and then practice the stretching exercises learned. They will be asked to track exercise electronically and on paper for 4 weeks. Participants will be compensated for participation.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of definite MS

* At least 18 years old
* Able to walk 25 feet independently with common assistive devices if needed
* Presence of spasticity by self-report interfering with usual daily activities
* Have an email account and be familiar with using it
* Willing to track daily exercise for 4 weeks
* Fluent in English

Exclusion Criteria:

Other medical or behavioral conditions that would limit participation or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda L Hugos, MS, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A Spasticity: Take Control | B Usual Care
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Spasticity: Take Control | B Usual Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.38 (12.79) | 52.83 (12.34) | 53.1 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: MS Walking Scale-12 (MSWS-12)
Description: The MSWS-12 is a clinically validated and reliable tool that is flexible and simple enough to use clinically and in research. It captures patients' perspectives on their ambulatory disability on the following: standing, ability to run, need for support, moving around the home, concentration needed to walk, walking speed, maintaining balance, climbing stairs, walking distance, effort needed to walk, ability to walk, and gait. It is simple to administer and responsive to changes in patient performance over time.
  Individual items are scored on a 5 point Likert scale: 1 (Not at all), 2 (A little), 3 (Moderately), 4 (Quite a bit), 5 (Extremely). A total score is generated and reported on a 0 to 100 scale by subtracting the minimum score possible (12) from the patient's score, dividing by the maximum score possible minus the minimum possible (60-12, or 48), and multiplying. Higher values represent a worse outcome and greater disability.
Time Frame: at average of 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Spasticity: Take Control | B Usual Care
Number analyzed (Participants) | 19 | 19
units on a scale | 72.6 (27.3) | 82.2 (30.8)
Statistical Analysis 1: Comparison: A Spasticity: Take Control vs B Usual Care; Test type: Superiority or Other; p = 0.84, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Timed 25 Foot Walk
Description: The time to walk 25 feet is strongly related to its ordinal counterpart the Ambulation Index (Spearman r=0.91) without the variability the ordinal scale reflects.
  The time is measured and recorded in seconds how long it takes for the participant to walk 25 feet.
Time Frame: at average of 4 months
Population: One subject was unable to complete this physical assessment at the visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | A Spasticity: Take Control | B Usual Care
Number analyzed (Participants) | 19 | 18
seconds | 7.6 (7) | 9.4 (10.4)
Statistical Analysis 1: Comparison: A Spasticity: Take Control vs B Usual Care; Test type: Superiority or Other; p = 0.738, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Timed up and go Test
Description: The Timed Up and Go (TUG) test measures the time in seconds it takes to get up from a chair, walk 10 feet, turn around and return to sit in the chair.
  The best score of the two attempts was analyzed.
Time Frame: at average of 4 months
Population: One subject was unable to complete this physical assessment at the visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | A Spasticity: Take Control | B Usual Care
Number analyzed (Participants) | 19 | 18
seconds | 11.23 (9.69) | 13.82 (13.51)
Statistical Analysis 1: Comparison: A Spasticity: Take Control vs B Usual Care; Test type: Superiority or Other; p = 0.8434, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: 2 Minute Walk Test
Description: The subject walks without assistance of another person for 2 minutes. The distance in feet the individual was able to walk in 2 minutes is then measured.
Time Frame: at average of 4 months
Population: One subject was unable to complete this physical assessment at the visit.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | A Spasticity: Take Control | B Usual Care
Number analyzed (Participants) | 19 | 18
feet | 462.8 (150.5) | 412.5 (158.7)
Statistical Analysis 1: Comparison: A Spasticity: Take Control vs B Usual Care; Test type: Superiority or Other; p = 0.638, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Modified Fatigue Impact Scale (MFIS)
Description: This self-report retrospective questionnaire measures fatigue symptoms. It consists of 21 items scored 0-4 for a total score between 0 and 84 and has a coefficient alpha of 0.81. Lower scores on the MFIS indicate less fatigue.
Time Frame: at average of 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Spasticity: Take Control | B Usual Care
Number analyzed (Participants) | 19 | 19
units on a scale | 41.1 (19.2) | 43.5 (20.8)
Statistical Analysis 1: Comparison: A Spasticity: Take Control vs B Usual Care; Test type: Superiority or Other; p = 0.492, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Multiple Sclerosis Impact Scale (MSIS-29)
Description: The MSIS-29 is designed to measure the physical and psychological impact of MS.
  Each subscale summed separately. No total calculated. Scores transformed to have a range of 0-100. Lower scores indicate less impact, higher scores indicate higher impact.
Time Frame: at average of 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Spasticity: Take Control | B Usual Care
Number analyzed (Participants) | 19 | 19
units on a scale
  MSIS-29 Physical | 45.6 (17.2) | 52.4 (19.2)
  MSIS-29 Psychological | 18.2 (7.6) | 20.6 (7.6)
Statistical Analysis 1: Comparison: A Spasticity: Take Control vs B Usual Care; This analysis refers to the physical component of the MSIS-29; Test type: Superiority or Other; p = 0.144, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: A Spasticity: Take Control vs B Usual Care; This refers to the psychological analysis for the MSIS-29; Test type: Superiority or Other; p = 0.953, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Spasticity Measured by the Modified Ashworth Scale
Description: The modified Ashworth Scale is a standard clinical and research method to quantify spasticity.
  Each of the 6 leg groups is given a scale of 0-4.
  0 - Normal. No increase in muscle tone.
  1. - Mild. Barely increased muscle tone. (catch)
  2. - Moderate. Moderately increased muscle tone that can be overcome and full range of motion is possible. (catch and resistance)
  3. - Severe. Severely increased muscle tone that is extremely difficult to overcome and full range of motion is not possible. (resistance and stop)
  4. - Contracted. All groups are summed for a total score for each side of the body. Higher scores indicate greater spasticity. Lowest possible score is a 0 whereas the highest possible score for each side is 24.
Time Frame: at average of 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Spasticity: Take Control | B Usual Care
Number analyzed (Participants) | 19 | 19
units on a scale | 10.8 (9.5) | 10.8 (9.3)
Statistical Analysis 1: Comparison: A Spasticity: Take Control vs B Usual Care; Test type: Superiority or Other; p = 0.915, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Multiple Sclerosis Spasticity Scale - 88 (MSSS-88)
Description: The modified MSSS-88 is a standardized self-report questionnaire to quantify subject's impact of the effects of spasticity.
  The 88 questions each have a possible score of 1-4. All questions are totaled for a final total scores. Higher scores indicate greater spasticity. The lowest score is 88 and the highest possible is 352.
Time Frame: at average of 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Spasticity: Take Control | B Usual Care
Number analyzed (Participants) | 19 | 19
units on a scale | 165.7 (53.3) | 192.4 (58.8)
Statistical Analysis 1: Comparison: A Spasticity: Take Control vs B Usual Care; Test type: Superiority or Other; p = 0.023, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Beck Depression Inventory II (BDI II)
Description: The BDI-II is a standardized self-report questionnaire to quantify depression.
  The BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. Answers to 21 questions added together. Higher scores indicate greater depression. Lowest possible score is a 0 whereas highest 63.
Time Frame: at average of 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Spasticity: Take Control | B Usual Care
Number analyzed (Participants) | 19 | 19
units on a scale | 9 (7.5) | 11.5 (8)
Statistical Analysis 1: Comparison: A Spasticity: Take Control vs B Usual Care; Test type: Superiority or Other; p = 0.11, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | A Spasticity: Take Control | B Usual Care
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 5/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Spasticity: Take Control (N=19) | B Usual Care (N=19)
Concussion (Nervous system disorders) | 0 (0) | 1 (1)
Leg spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
Broken arm resulting from fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pain and bruising from fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Increase in urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes